CLINICAL TRIAL: NCT07018076
Title: Candidate Clinical Correlate of Prognostic Outcome for TB Study
Acronym: C3PO
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Irvine (Other); University of Colorado, Denver (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: U01AI152087-05S1 (NIH); U01AI152087-05S1 (NIH)
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Global Health; Diagnostics
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: RS ratio — We will evaluate the non-culture, sputum-based assay RS ratio, which measures ongoing Mycobacterium tuberculosis activity by quantifying the abundance of precursor rRNA relative to mature rRNA (an indicator of active rRNA synthesis).
Diagnostic Test: Blood-based host immune response assays — We will evaluate blood-based assays measuring host immune response parameters for predicting mycobacterial activity.

SUMMARY:
As part of the ongoing efforts within the Rapid Research in Diagnostics Development for TB Network (R2D2 TB Network) study, the Candidate Clinical Correlate as Prognostic Outcome for TB (C3PO) study serves as a supplement aimed at evaluating predictors and novel biomarkers of recurrent TB among TB survivors. Current tools for predicting TB recurrence risk are suboptimal, limiting the ability to assess new TB treatment regimens effectively. Identifying accurate sputum- or blood-based biomarkers for recurrence risk could significantly improve the efficiency and informativeness of Phase 2 and 3 clinical trials.

DETAILED DESCRIPTION:
The Candidate Clinical Correlate as Prognostic Outcome for TB Study (C3PO) supplements the ongoing Rapid Research in Diagnostics Development for TB Network (R2D2 TB Network) study by identifying and accelerating novel TB diagnostics at various stages of development and across different use cases. There is an urgent need for treatments that can cure all forms of TB more quickly. However, the development of new, shorter, and more effective antibiotic regimens is hindered by the limitations of current methods used to assess treatment effectiveness in TB drug trials. The standard pharmacodynamic (PD) marker-sputum culture-does not predict clinical outcomes well, fails to detect residual Mycobacterium tuberculosis that causes relapse, and takes 6-8 weeks to provide results. New PD markers that more accurately predict clinical outcomes would help de-risk clinical trials and ensure that only the most effective new regimens move forward. C3PO aims to evaluate non-culture PD markers in predicting recurrent TB among patients who have completed the global standard HRZE regimen for drug-susceptible pulmonary TB under routine programmatic settings.

ELIGIBILITY:
Inclusion Criteria:

1. . individuals age ≥ 12 years;
2. . have completed treatment for drug-susceptible tuberculosis with the standard 6-month regimen of isoniazid, rifampin, pyrazinamide, and ethambutol (HRZE).

Exclusion Criteria:

1. completed treatment for drug-susceptible tuberculosis >14 days prior to screening/enrollment;
2. routinely taking any medication with anti-mycobacterial activity (including fluoroquinolones) for any reason not related to tuberculosis treatment within the last 14 days;
3. unwilling to provide informed consent or return for study follow-up visits.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of individuals receiving programmatic treatment for drug-sensitive tuberculosis (TB) at participating outpatient TB clinics in Uganda and Vietnam. Eligible participants will be selected from among TB patients actively receiving care at these clinical sites.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Recurrent tuberculosis (TB) | 1 year
  Recurrent tuberculosis (TB), defined as a new episode of microbiologically confirmed TB occurring after completion of treatment for a prior drug-sensitive TB episode. Recurrence will be identified through routine study visits during the one year follow-up, with microbiological confirmation based on sputum mycobacterial culture.
Prognostic accuracy of novel biomarkers in predicting recurrent TB | 1 year
  We will evaluate the ability of selected novel biomarkers to predict recurrent TB using the following metrics:
  Area Under the Curve (AUC): Measures the overall discriminatory ability of the biomarkers to distinguish between individuals who will and will not experience recurrent TB.
  Sensitivity and Specificity: Sensitivity indicates how accurately the biomarkers identify individuals who will develop recurrent TB, while specificity reflects how well they identify those who will not.
  Positive Predictive Value (PPV) and Negative Predictive Value (NPV): PPV represents the proportion of individuals with a positive biomarker result who actually develop recurrent TB, while NPV reflects the proportion with a negative result who remain recurrence-free.
  Kappa Statistic: Assesses the agreement between predicted outcomes based on the biomarkers and the actual observed outcomes, accounting for agreement occurring by chance.

CONTACTS AND LOCATIONS:
Overall Officials: Adithya Cattamanchi, MD, Principal Investigator — University of California San Francisco; University of California Irvine
Locations (3):
- Uganda (2):
  - Kisenyi Health Center, Kampala
  - Mulago Outpatient Department, Kampala
- Hanoi Lung Hospital, Outpatient departments, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] STREPTOMYCIN treatment of pulmonary tuberculosis. Br Med J. 1948 Oct 30;2(4582):769-82. No abstract available. PMID 18890300
- [Background] Sharma M, Nduba V, Njagi LN, Murithi W, Mwongera Z, Hawn TR, Patel SN, Horne DJ. TBscreen: A passive cough classifier for tuberculosis screening with a controlled dataset. Sci Adv. 2024 Jan 5;10(1):eadi0282. doi: 10.1126/sciadv.adi0282. Epub 2024 Jan 3. PMID 38170773
- [Background] Phillips PPJ, Mendel CM, Nunn AJ, McHugh TD, Crook AM, Hunt R, Bateson A, Gillespie SH. A comparison of liquid and solid culture for determining relapse and durable cure in phase III TB trials for new regimens. BMC Med. 2017 Nov 24;15(1):207. doi: 10.1186/s12916-017-0955-9. PMID 29169355
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Background] Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall GL, Culver BH, Enright PL, Hankinson JL, Ip MS, Zheng J, Stocks J; ERS Global Lung Function Initiative. Multi-ethnic reference values for spirometry for the 3-95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012 Dec;40(6):1324-43. doi: 10.1183/09031936.00080312. Epub 2012 Jun 27. PMID 22743675
- [Background] Kurbatova EV, Phillips PPJ, Dorman SE, Sizemore EE, Bryant KE, Purfield AE, Ricaldi J, Brown NE, Johnson JL, Wallis CL, Akol JP, Ocheretina O, Van Hung N, Mayanja-Kizza H, Lourens M, Dawson R, Nhung NV, Pierre S, Musodza Y, Shenje J, Badal-Faesen S, Vilbrun SC, Waja Z, Peddareddy L, Scott NA, Yuan Y, Goldberg SV, Swindells S, Chaisson RE, Nahid P. A Standardized Approach for Collection of Objective Data to Support Outcome Determination for Late-Phase Tuberculosis Clinical Trials. Am J Respir Crit Care Med. 2023 May 15;207(10):1376-1382. doi: 10.1164/rccm.202206-1118OC. PMID 36790881
- [Background] Horne DJ, Royce SE, Gooze L, Narita M, Hopewell PC, Nahid P, Steingart KR. Sputum monitoring during tuberculosis treatment for predicting outcome: systematic review and meta-analysis. Lancet Infect Dis. 2010 Jun;10(6):387-94. doi: 10.1016/S1473-3099(10)70071-2. PMID 20510279
- [Background] Imperial MZ, Phillips PPJ, Nahid P, Savic RM. Precision-Enhancing Risk Stratification Tools for Selecting Optimal Treatment Durations in Tuberculosis Clinical Trials. Am J Respir Crit Care Med. 2021 Nov 1;204(9):1086-1096. doi: 10.1164/rccm.202101-0117OC. PMID 34346856
- [Background] Gupta-Wright A, den Boon S, MacLean EL, Cirillo D, Cobelens F, Gillespie SH, Kohli M, Ruhwald M, Savic R, Brigden G, Gidado M, Goletti D, Hanna D, Hasan R, Hewison C, Koura KG, Lienhardt C, Lungu P, McHugh TD, McKenna L, Scott C, Scriba T, Sekaggya-Wiltshire C, Kasaeva T, Zignol M, Denkinger CM, Falzon D. Target product profiles: tests for tuberculosis treatment monitoring and optimization. Bull World Health Organ. 2023 Nov 1;101(11):730-737. doi: 10.2471/BLT.23.290901. Epub 2023 Oct 4. PMID 37961060
- [Background] FDA-NIH Biomarker Working Group. BEST (Biomarkers, EndpointS, and other Tools) Resource [Internet]. Silver Spring (MD): Food and Drug Administration (US); 2016-. Available from http://www.ncbi.nlm.nih.gov/books/NBK326791/ PMID 27010052
- [Background] MacLean EL, Zimmer AJ, den Boon S, Gupta-Wright A, Cirillo DM, Cobelens F, Gillespie SH, Nahid P, Phillips PP, Ruhwald M, Denkinger CM. Tuberculosis treatment monitoring tests during routine practice: study design guidance. Clin Microbiol Infect. 2024 Apr;30(4):481-488. doi: 10.1016/j.cmi.2023.12.027. Epub 2024 Jan 3. PMID 38182047
- [Background] Evangelopoulos D, Shoen CM, Honeyborne I, Clark S, Williams A, Mukamolova GV, Cynamon MH, McHugh TD. Culture-Free Enumeration of Mycobacterium tuberculosis in Mouse Tissues Using the Molecular Bacterial Load Assay for Preclinical Drug Development. Microorganisms. 2022 Feb 17;10(2):460. doi: 10.3390/microorganisms10020460. PMID 35208914
- [Background] MCCUNE RM Jr, MCDERMOTT W, TOMPSETT R. The fate of Mycobacterium tuberculosis in mouse tissues as determined by the microbial enumeration technique. II. The conversion of tuberculous infection to the latent state by the administration of pyrazinamide and a companion drug. J Exp Med. 1956 Nov 1;104(5):763-802. doi: 10.1084/jem.104.5.763. PMID 13367342
- [Background] Mukamolova GV, Turapov O, Malkin J, Woltmann G, Barer MR. Resuscitation-promoting factors reveal an occult population of tubercle Bacilli in Sputum. Am J Respir Crit Care Med. 2010 Jan 15;181(2):174-80. doi: 10.1164/rccm.200905-0661OC. Epub 2009 Oct 29. PMID 19875686
- [Background] Dorman SE, Nahid P, Kurbatova EV, Phillips PPJ, Bryant K, Dooley KE, Engle M, Goldberg SV, Phan HTT, Hakim J, Johnson JL, Lourens M, Martinson NA, Muzanyi G, Narunsky K, Nerette S, Nguyen NV, Pham TH, Pierre S, Purfield AE, Samaneka W, Savic RM, Sanne I, Scott NA, Shenje J, Sizemore E, Vernon A, Waja Z, Weiner M, Swindells S, Chaisson RE; AIDS Clinical Trials Group; Tuberculosis Trials Consortium. Four-Month Rifapentine Regimens with or without Moxifloxacin for Tuberculosis. N Engl J Med. 2021 May 6;384(18):1705-1718. doi: 10.1056/NEJMoa2033400. PMID 33951360
- [Background] Gillespie SH, Crook AM, McHugh TD, Mendel CM, Meredith SK, Murray SR, Pappas F, Phillips PP, Nunn AJ; REMoxTB Consortium. Four-month moxifloxacin-based regimens for drug-sensitive tuberculosis. N Engl J Med. 2014 Oct 23;371(17):1577-87. doi: 10.1056/NEJMoa1407426. Epub 2014 Sep 7. PMID 25196020
- [Background] Nahid P, Dorman SE, Alipanah N, Barry PM, Brozek JL, Cattamanchi A, Chaisson LH, Chaisson RE, Daley CL, Grzemska M, Higashi JM, Ho CS, Hopewell PC, Keshavjee SA, Lienhardt C, Menzies R, Merrifield C, Narita M, O'Brien R, Peloquin CA, Raftery A, Saukkonen J, Schaaf HS, Sotgiu G, Starke JR, Migliori GB, Vernon A. Official American Thoracic Society/Centers for Disease Control and Prevention/Infectious Diseases Society of America Clinical Practice Guidelines: Treatment of Drug-Susceptible Tuberculosis. Clin Infect Dis. 2016 Oct 1;63(7):e147-e195. doi: 10.1093/cid/ciw376. Epub 2016 Aug 10. PMID 27516382
- [Background] Walter ND, Born SEM, Robertson GT, Reichlen M, Dide-Agossou C, Ektnitphong VA, Rossmassler K, Ramey ME, Bauman AA, Ozols V, Bearrows SC, Schoolnik G, Dolganov G, Garcia B, Musisi E, Worodria W, Huang L, Davis JL, Nguyen NV, Nguyen HV, Nguyen ATV, Phan H, Wilusz C, Podell BK, Sanoussi ND, de Jong BC, Merle CS, Affolabi D, McIlleron H, Garcia-Cremades M, Maidji E, Eshun-Wilson F, Aguilar-Rodriguez B, Karthikeyan D, Mdluli K, Bansbach C, Lenaerts AJ, Savic RM, Nahid P, Vasquez JJ, Voskuil MI. Mycobacterium tuberculosis precursor rRNA as a measure of treatment-shortening activity of drugs and regimens. Nat Commun. 2021 May 18;12(1):2899. doi: 10.1038/s41467-021-22833-6. PMID 34006838
- [Background] Linh NN, Viney K, Gegia M, Falzon D, Glaziou P, Floyd K, Timimi H, Ismail N, Zignol M, Kasaeva T, Mirzayev F. World Health Organization treatment outcome definitions for tuberculosis: 2021 update. Eur Respir J. 2021 Aug 19;58(2):2100804. doi: 10.1183/13993003.00804-2021. Print 2021 Aug. No abstract available. PMID 34413124
- [Background] Phillips PP, Mendel CM, Burger DA, Crook AM, Nunn AJ, Dawson R, Diacon AH, Gillespie SH. Limited role of culture conversion for decision-making in individual patient care and for advancing novel regimens to confirmatory clinical trials. BMC Med. 2016 Feb 4;14:19. doi: 10.1186/s12916-016-0565-y. PMID 26847437
- [Background] Dooley KE, Phillips PP, Nahid P, Hoelscher M. Challenges in the clinical assessment of novel tuberculosis drugs. Adv Drug Deliv Rev. 2016 Jul 1;102:116-22. doi: 10.1016/j.addr.2016.01.014. Epub 2016 Jan 28. PMID 26827911
- [Background] Ivanova O, Hoffmann VS, Lange C, Hoelscher M, Rachow A. Post-tuberculosis lung impairment: systematic review and meta-analysis of spirometry data from 14 621 people. Eur Respir Rev. 2023 Apr 19;32(168):220221. doi: 10.1183/16000617.0221-2022. Print 2023 Jun 30. PMID 37076175
- [Background] Dide-Agossou C, Bauman AA, Ramey ME, Rossmassler K, Al Mubarak R, Pauly S, Voskuil MI, Garcia-Cremades M, Savic RM, Nahid P, Moore CM, Tasneen R, Nuermberger EL, Robertson GT, Walter ND. Combination of Mycobacterium tuberculosis RS Ratio and CFU Improves the Ability of Murine Efficacy Experiments to Distinguish between Drug Treatments. Antimicrob Agents Chemother. 2022 Apr 19;66(4):e0231021. doi: 10.1128/aac.02310-21. Epub 2022 Mar 21. PMID 35311519